CLINICAL TRIAL: NCT06849011
Title: Development and Validation of a Prognostic Prediction Model for Adverse Outcomes in Neurocritical Patients Receiving Enteral Nutrition Based on Key Inflammatory and Metabolic Markers
Brief Title: Inflammatory and Metabolic Prognostic Assessment in Critically Ill Neurological Patients
Acronym: IMPACT-NEURO
Status: Not yet recruiting | Type: Observational
Sponsor: Yan Zhang (Other)
Responsible Party: Sponsor-Investigator, Yan Zhang, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: xwzc202500102
Record Dates: First submitted 2025-02-12; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke Acute; Encephalitis; Non-traumatic Brain Injury
Keywords: enteral nutrition; adverse prognosis; prediction model; non-traumatic severe brain injury
MeSH Terms: conditions — Stroke; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and gastric juice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- mild Inflammation & Metabolic dysfunction: First, a predictive model for poor prognosis is constructed through screening of independent variables after data collection. Then, stratified analysis is conducted with inflammatory markers such as C-reactive protein and interleukin-6, and metabolic markers such as blood glucose and insulin dosage.
- Moderate Inflammation & Metabolic Dysregulation: First, a predictive model for poor prognosis is constructed through screening of independent variables after data collection. Then, stratified analysis is conducted with inflammatory markers such as C-reactive protein and interleukin-6, and metabolic markers such as blood glucose and insulin dosage.
- High Inflammation & Severe Metabolic Dysregulation: First, a predictive model for poor prognosis is constructed through screening of independent variables after data collection. Then, stratified analysis is conducted with inflammatory markers such as C-reactive protein and interleukin-6, and metabolic markers such as blood glucose and insulin dosage.
- Peptide-Based Nutrition: Select patients who received peptide-based formulas from the entire database for poor prognosis analysis.
- Whole Protein Nutrition: Select patients who received whole protein formulas from the database for poor prognosis analysis.

SUMMARY:
The study aims to develop and validate a prognostic prediction model for adverse outcomes in neurocritical patients receiving enteral nutrition based on key inflammatory and metabolic markers. This model will serve as a clinical tool to help physicians identify high-risk patients and guide individualized nutritional support strategies.

DETAILED DESCRIPTION:
A multi-center, prospective case data collection study will be conducted across 19 tertiary hospitals in China. Based on this, a predictive assessment model for poor prognosis in neurocritically ill patients receiving enteral nutrition support will be developed and validated, using key inflammatory and metabolic markers. During the data collection process, comprehensive clinical information will be extracted, including patient demographic data, clinical indicators, and hematological markers. By conducting in-depth analysis and processing of this vast and detailed clinical and laboratory data, a nomogram for predicting poor prognosis in neurocritical care patients receiving enteral nutrition support will be constructed using statistical methods and data analysis techniques in R. Once the model is built, it will undergo rigorous validation on an independent external dataset to ensure its accuracy and reliability. The goal is to create a precise assessment tool for clinicians, helping them to quickly and accurately identify high-nutritional-risk patients, thereby providing a solid scientific foundation for the formulation of individualized nutrition support strategies, ultimately improving the prognosis of neurocritical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, no gender restrictions.
2. Within 7 days of disease onset and expected NICU stay of at least 7 days.
3. Eligible for enrollment within 24 hours of NICU admission, with enteral nutrition (EN) initiated and continued for at least 7 days.
4. Non-traumatic severe brain injury patients (including cerebrovascular disease and encephalitis) with a Glasgow Coma Scale (GCS) score ≤12.
5. NRS 2002 score ≥3.
6. Kuwata drinking test ≥ grade 3.
7. Acute Gastrointestinal Injury (AGI) grade 1 or 2.
8. Signed informed consent obtained from the patient or their legal representative.

Exclusion Criteria:

1. Severe malnutrition prior to admission, defined as BMI < 16 kg/m².
2. Pregnant or lactating women.
3. Receiving hypothermia treatment or core body temperature < 36°C.
4. End-stage disease with an expected survival time of < 48 hours, or severe dysfunction of the heart, lungs, or other vital organs, leading to hemodynamic instability.
5. Malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of critically ill neurocritical patients in the acute phase who are receiving enteral nutrition (EN) treatment in the Neurocritical Care Unit (NICU).
Sampling Method: Non-Probability Sample
Enrollment: 1185 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at Day 28 of enteral nutrition therapy | From enrollment to 28 days after the initiation of enteral nutrition

SECONDARY OUTCOMES:
Nutritional goal achievement rate at Day 3 (caloric and protein intake reaching 70%-100% of calculated target) | At Day 3 after the initiation of enteral nutrition
Adverse outcome rate at Day 90 (defined as a Modified Rankin Scale score ≥ 3) | At Day 90 after the initiation of enteral nutrition
Incidence of infectious complications within 14 days (including pneumonia, urinary tract infections, bloodstream infections, skin infections, and Clostridium difficile infections) | Within 14 days after the initiation of enteral nutrition
Gastrointestinal intolerance within 14 days (gastric residual volume > 200 mL, nausea, vomiting, bloating, diarrhea) | Within 14 days after the initiation of enteral nutrition
  The gastric residual volume is assessed every 4 hours by the nurse through aspiration via the nasogastric tube. Other clinical manifestations such as nausea, vomiting, bloating, and diarrhea are assessed through daily observation by the attending physician.
Incidence of gastrointestinal bleeding within 14 days (gastric occult blood, fecal occult blood, hematemesis, melena, hematochezia) | Within 14 days after the initiation of enteral nutrition
Number of days with random blood glucose > 10 mmol/L within 14 days | Within 14 days after the initiation of enteral nutrition
Average daily insulin requirement within 14 days | Within 14 days after the initiation of enteral nutrition
Incidence of hypophosphatemia within 3 days | Within 3 days after the initiation of enteral nutrition
Duration of mechanical ventilation within 14 days | Within 14 days after the initiation of enteral nutrition
Length of NICU stay | From enrollment to discharge from the NICU, up to 1 year.
Total hospital stay duration | From enrollment to discharge, up to 1 year.
90-day readmission rate post-discharge | Within 90 days after discharge

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing Hui People's Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - You'anmen Hospital, Beijing, Beijing Municipality
  - The Ninth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The 940th Hospital of Joint Logistics Support Force of Chinese PLA, Lanzhou, Gansu
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Tangshan People's Hospital, Tangshan, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Heibei
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Jilin, Jilin
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The 960th Hospital of Joint Logistics Support Force of Chinese PLA, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared. Available data includes demographic information, clinical characteristics, laboratory results, and outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon reasonable request from 6 months after study completion to 3 years post-publication.
Access Criteria: Access will be granted to qualified researchers upon reasonable request through a formal data-sharing agreement.